CLINICAL TRIAL: NCT05692193
Title: The Effect Of Pre-Surgery Paın Educatıon On Postoperatıve Paın And Comfort In Anorectal Dıseases
Brief Title: The Effect of Pain Education on Pain and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Muhsin UYSAL, Surgical Nurse, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022/11
Record Dates: First submitted 2023-01-06; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative
Keywords: Anorectal diseases; pain; confort; Pain education
MeSH Terms: conditions — Pain, Postoperative; Rectal Diseases; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): * A 'Patient Pain Education Brochure', which was prepared the day before the surgery, was given, and at the same time, the training was given verbally and in writing for an average of 20-30 minutes in the patient's own room.
  * Vital sessions and pain assessment were performed during admission to the ward before the training.
  * Pain was evaluated together with the patient's vital signs at the 15th, 30th, 45th, 60th minutes, 2nd, 4th, 6th, 12th, and 24th hours after the surgery.
  * Comfort assessment was performed at the 24th hour after surgery.
  Interventions: Behavioral: pain education
- control group (No Intervention): * One day before the operation, vital signs and pain were evaluated during hospitalization.
  * Pain was evaluated together with the patient's vital signs at the 15th, 30th, 45th, 60th minutes, 2nd, 4th, 6th, 12th, and 24th hours after the surgery.
  * Comfort assessment was performed at the 24th hour after surgery.

INTERVENTIONS:
Behavioral: pain education — Pain education was given to the experimental group for 20-30 minutes on the day of hospitalization.
  Arms: experimental group

SUMMARY:
The study was planned as quasi-experimental to determine the effect of pain training given to patients who will undergo surgery for anorectal diseases on postoperative pain and comfort. The research was carried out in Istanbul Taksim Training and Research Hospital General Surgery Clinic between November 2021 and November 2022. Data were collected with the "Patient Introduction Education Leaflet", "Patient Pain Education Leaflet", "Numeric Pain Scale", "Brief Pain Inventory" and "Perianesthesia Comfort Scale". The data were analyzed with appropriate statistical methods using the SPSS 25.0 package program.

In the study, the difference between the groups in terms of demographic characteristics and life histories of the patients was insignificant and showed a homogeneous distribution (p>0.05). When the measurements of the patients in the experimental and control groups were compared; It was determined that the patients in the experimental group had lower pulse, blood pressure, respiratory rate and body temperature, and the mean SPO2 was higher than the patients in the control group (p<0.05). When the evaluations between the groups are examined; It was found that the mean pain scores evaluated with the Numerical Pain Scale and Brief Pain Inventory scales in the patients included in the experimental group were lower than the patients included in the control group; The comfort level evaluated with the Perianesthesia Comfort Scale was found to be higher in the experimental group than in the control group (p<0.05).

Hypothesis 1: Pain education given to experimental group patients who will undergo surgery for anorectal diseases has an effect on postoperative pain.

Hypothesis 2: Pain education given to patients in the experimental group who will undergo surgery for anorectal diseases has an effect on the comfort level after surgery.

DETAILED DESCRIPTION:
Type of research: The research was planned as quasi-experimental. Location: The study is planned to be carried out with patients who were planned for anorectal surgery and hospitalized in Taksim Training and Research Hospital General Surgery Clinic in Beyoğlu district of Istanbul.

Population, sampling method and number: The population of the study will consist of patients who will undergo hemorrhoid, anal abscess, anal fissure or anal fistula surgery in the General Surgery Clinic in Taksim Training and Research Hospital in Istanbul.

There are different methods to determine the sample size in the literature. In this study, the sample size for repeated ANOVA measures will be calculated using the medium effect size standardized by Cohen. Sample calculation will be done with G-power 3.1 package program. The sample of the study will be determined as at least 36 patients in each of the case and control groups, with an effect size of 0.25 and a power of 0.90. Considering that there may be case losses due to any reason and cases that can be excluded from the sample in terms of homogeneity of the groups, it will be planned to include 40 patients in the study and control groups by increasing it by 10%. Being over 18 years old, being literate, having surgery for anorectal diseases, having surgery under spinal anesthesia and volunteering to participate in the study will be determined as inclusion criteria.

Dependent Variables: Heart rate, respiratory rate, oxygen saturation, body temperature, blood pressure, pain score constitute the dependent variables.

Independent Variables: Gender, age, weight, height, occupation, income level and previous surgeries constitute the independent variables.

Statistical analysis methods to be used: The data obtained from the research will be transferred to the electronic environment and evaluated in the SPSS 25.0 package program. Number, percentage, mean and standard deviation will be used as descriptive statistical methods in the evaluation of the data. Before the data analysis, normality test will be done to test the compliance with the parametric test methods. In order to test the normal distribution condition, Kolmogorov Smirnov Z test will be applied. Chi-square and Fisher's exact tests will be applied to determine the homogeneity of the groups. In line with the results, the data will be analyzed with the related tests. The findings will be evaluated at the 95% confidence interval and at the 5% significance level.

In order to obtain the data of the study, "Patient Identification Form", "Patient Pain Education Brochure", "Numerical Pain Scale" , "Short Pain Inventory" prepared by the researcher by scanning the literature., "Perianesthesia Comfort Scale" will be used. In the quasi-experimental study, the patients will be divided into two groups as the experimental and control group by simple random method. The patients in the experimental group will be given the "Patient Pain Education Brochure" prepared one day before the surgery, taking into account the individual and pandemic measures, and at the same time, the training will be given verbally and in writing for an average of 20-30 minutes in the patient's own room. With the patient's vital signs at the time of admission to the ward before the training, immediately after the training and at the 15th, 30th, 45th, 60th minutes, 2nd, 4th, 6th, 12th, and 24th hours after the operation, to the intervention group that was trained. "Numerical Pain Scale", "Brief Pain Inventory" , "Perianesthesia Comfort Scale" will be applied at the 24th hour. Patients in the control group will not be given pain training, and vital signs of the patient during their hospitalization, one day before the operation and at the 15th, 30th, 45th, 60th minutes, 2nd, 4th, 6th, 12th, 24th hours after the operation. "Numerical Pain Scale" , "Brief Pain Inventory" , "Perianesthesia Comfort Scale" will be applied at the 24th hour. The patients will be informed about the purpose of the research, benefits, duration of education, scale forms and evaluation periods by the researcher, and an "Informed Consent" will be obtained by explaining that their individual rights will be protected and their personal information will be kept confidential. The patient education brochure will be submitted to the expert opinion of 10 people for content evaluation. The brochure will be finalized according to the suggestions of the experts. The prepared training will be applied to 10 patients for content and language validity.

ELIGIBILITY:
Inclusion Criteria:

- Being over 18 years old, literate, having surgery for anorectal diseases, having surgery under spinal anesthesia and volunteering to participate in the research.

Exclusion Criteria:

* using analgesia, mentally ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Pain score | Hospitalization day (0. minute)
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 15 minutes after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 30 minutes after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 45 minutes after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 60 minutes after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 120 minutes after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 4. hours after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 6. hours after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 12. hours after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.
Pain Score | 24. hours after surgery
  Pain intensity is measured as a numerical pain scale (0 = no pain, 10 = excruciating pain). The degree of pain expressed by the individual measures the general activity state caused by the pain in the last 24 hours, emotional state, relationships with other people, ability to walk, exercise, sleep, and enjoyment of life. Each item is evaluated as a numerical pain scale from 0 to 10 (0 = not affected at all, 10 = completely affected). The patient can mark the area where he feels pain on the picture, which method or drugs are used to provide analgesia, and the level of describing the pain in the last 24 hours is evaluated with percentages. In the brief pain inventory, pain is defined as 1-4 mild pain, 5-6 moderate and 7-10 severe pain.

SECONDARY OUTCOMES:
Comfort level | 24. hours after surgery
  The Perianesthesia Comfort Scale is a one-dimensional scale consisting of 24 items that reflects the individual's thought process before and after surgery and questions his feelings. Each statement in the scale is scored on a Likert type ranging from 1 to 6, from 'strongly disagree' to 'strongly agree'. Accordingly, a high score (6 points) for positive items indicates high comfort, a low score (1 point) indicates low comfort, and a low score (1 point) for negative items indicates high comfort, and a high score (6 points) indicates low comfort. The highest total score that can be obtained on the scale is 144, and the lowest total score is 24. The average value is determined by dividing the total score obtained by the number of scale items, and the result is indicated in the 1-6 distribution. A low score indicates poor comfort, while a high score indicates good comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Muhsin Uysal, Researcher, Principal Investigator — Istanbul Taksim Training and Research Hospital
Locations (1):
- Home, Istanbul, Üskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No